CLINICAL TRIAL: NCT07163182
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of CHF6467 After Single and Repeated Ascending Doses by Intranasal Route in Healthy Adult Subjects
Brief Title: Evaluation of Safety, Side Effects and How the Drug CHF6467 Administered Via Intranasal Route is Absorbed, Modified and Removed in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-06467AC1-02; 2025-521455-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-24; First posted 2025-09-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: Single Ascending Dose; Multiple Ascending Dose; Intranasal; Cerebrospinal fluid
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: Part 1 - SAD (single ascending dose): Randomised, double-blind, placebo-controlled, single-dose escalation, parallel-group design in healthy volunteers (HVs).
  Part 2 - MAD (multiple ascending dose): Randomised, double-blind, placebo-controlled, repeated-dose escalation, parallel-group design in HVs.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigational Medicinal Product is blinded for the participant, the investigators and the Sponsor. At site an unblind pharmacist is foreseen to prepare the Investigational Medicinal Product and an unblinded Clinical Research Associate will check the documents of the Investigational Medicinal Product preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Treatment (Active Comparator): Intranasal (IN) CHF6467
  Interventions: Biological: CHF6467 Part 1 (SAD); Biological: CHF6467 Part 2 (MAD)
- Reference Treatment (Placebo Comparator): Intranasal (IN) placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CHF6467 Part 1 (SAD) — Intranasal administration of single ascending doses of CHF6467 in 4 different cohorts
  Arms: Test Treatment
Biological: CHF6467 Part 2 (MAD) — Intranasal administration of multiple ascending doses of CHF6467 in 3 different cohorts
  Arms: Test Treatment
Drug: Placebo — Intranasal administration of matched-placebo of CHF6467 in Part 1 and Part 2
  Arms: Reference Treatment

SUMMARY:
A clinical trial to investigate the safety and tolerability of single and multiple intranasal (through the nose) dosing with the study drug CHF6467 in 68 healthy adult subjects.

The study will investigate also how CHF6467 moves and behaves in the blood and in the fluid around the brain and spinal cord (cerebrospinal fluid) and if the drug CHF6467 causes an immune response by looking for specific molecules, called antibodies that may form against it.

The study will be divided into two parts - Part 1 (testing single ascending doses of the study drug, SAD, lasting 4 days) and Part 2 (testing repeated or multiple ascending doses of the study drug, MAD, lasting 11 days).

Each part of the study consists of a screening period, when eligible healthy volunteers will be selected, a treatment period, during which the study drug administration will take place and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedures;
2. Willingness and ability to understand the risks involved and to understand and comply with the study procedures;
3. Healthy male and female subjects, aged 18-55 years inclusive at screening;
4. Weight ≥ 50 kg and <85 kg and Body Mass Index (BMI) between 18.0 and 30.0 kg/m² inclusive at screening and on Day -1;
5. Non-smoker or ex-smoker who smoked less than 5 pack years (Pack years = the number of cigarette packs per day times the number of years) and stopped smoking at least 1 year prior to screening;
6. Good physical condition and mental status determined by the Investigator, based on the subject's medical history and general clinical examination at screening and Day -1;
7. Vital signs within normal limits at screening and at Day-1: 60 mmHg ≤ diastolic blood pressure (DBP) ≤ 89 mmHg, 90 mmHg ≤ systolic blood pressure (SBP) ≤ 139 mmHg (three measures performed after at least 5 minutes of resting; the mean value must be within the defined range). Axillary body temperature of 35.5-37.0º Celsius inclusive;
8. Bedside 12-lead electrocardiogram (ECG) considered as normal (45 bpm ≤ heart rate [HR] ≤ 100 bpm, 120 ms ≤ PR interval [PR] ≤ 210 ms, QRS interval [QRS] ≤ 120 ms, QT interval [QT] corrected using Fridericia's formula [QTcF] ≤ 450 ms for males and ≤ 470 ms for females) at screening visit and Day -1; the mean value of three measurements must be within the range.
9. Males fulfilling one of the following criteria:

   1. Males with pregnant or non-pregnant women of childbearing potential (WOCBP) partners: they must be willing to use male condom from the signature of the informed consent and until the follow-up visit or
   2. Non-fertile male subjects (contraception is not required in this case) or
   3. Males with partner not of childbearing potential (contraception is not required in this case);
10. Female subjects fulfilling one of the following criteria:

    1. Women of non-childbearing potential (WOCBP) defined as physiologically incapable of becoming pregnant (i.e., post-menopausal or permanently sterile). Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per Investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone (FSH) levels (according to local laboratory ranges);
    2. WOCBP fulfilling one of the following criteria:

    i. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method preferably with low user dependency from the signature of the informed consent and until the follow-up visit; or ii. WOCBP with non-fertile male partners (contraception is not required in this case).

Exclusion Criteria:

1. The subject has taken non-permitted concomitant medications in the predefined period prior to screening or prior to randomisation or is expected to take non-permitted concomitant medications during the study;
2. Participation to investigational study: subjects who have received any investigational drug within the 30 days (60 days for biologics) or a more appropriate time as determined by the Investigator (e.g. approximately 5 half-lives of the investigational drug whatever is longer);
3. Significant nasal congestion or signs of nasal damage, bleeding, excoriation or ulceration at physical examination at screening or Day -1;
4. History of frequent nosebleeds;
5. Any ongoing acute (e.g. non-allergic rhinitis) or chronic (e.g. chronic rhinosinusitis or chronic purulent postnasal drip) condition of the nasal cavity, or clinically significant physical finding (e.g. nasal polyps, nasal structural abnormalities, nasal trauma, severe nasal septal deviation) which, in the opinion of the Investigator, can interfere with the administration or absorption of the study medication. Subjects with recent upper respiratory tract infections will be allowed in the study only if their nasal symptoms have been completely resolved for more than 2 weeks prior to screening;
6. Clinically significant abnormal 24-hour Holter at screening;
7. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic or psychiatric disorder that may interfere with successful completion of this protocol, any known malignancies, or any condition that in Investigator's opinion may pose the subject at risk from participating in the study;
8. Any clinically relevant abnormal laboratory value at screening or Day -1suggesting an undiagnosed condition that requires further clinical investigation or may impact the safety of the subject or the evaluation of the study results according to the Investigator's judgement; Note: In case of abnormal laboratory values that could indicate a temporary condition, the test can be repeated once before randomisation;
9. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test. Serum pregnancy test to be performed at screening and urine pregnancy test to be performed at Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Adverse Drug Reactions (ADRs) | From screening (3 to 21 days prior to Day 1) to the last follow-up visit (29 ±3 days after Day 1 for Part 1; 85 ±3 days after Day 1 for Part 2)
  Number of events and number and percentage of subjects experiencing treatment-emergent AEs (TEAEs), treatment-emergent ADRs, serious TEAEs, non-serious TEAEs, severe TEAEs, TEAEs leading to discontinuation of study treatment and TEAEs leading to death
Vital signs: heart rate (HR) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Mean absolute value
Vital signs: body temperature (BT) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after randomisation for Part 1; between 7 and 14 days after last administration for Part 2)
  Mean absolute value
Vital signs: systolic blood pressure (SBP), diastolic blood pressure (DBP) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  * Mean absolute value
  * Mean change from baseline
Bedside 12-lead ECG intervals (HR, PR, QRS, QT, QTcF) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Mean absolute value
Bedside 12-lead ECG intervals (HR, PR, QRS, QT, QTcF) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Mean change from baseline
Bedside 12-lead ECG intervals (HR, PR, QRS, QT, QTcF) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Mean difference vs. placebo in change from baseline
Bedside 12-lead ECG intervals (HR, PR, QRS, QT, QTcF) | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Number and percentage of subjects with:
  * QTcF > 450 ms, > 480 ms and > 500 ms;
  * Change from baseline in QTcF > 30 ms and > 60 ms
12-lead ECG parameters extracted from Holter (HR, PR, QRS, QTcF and QT) | From Day 1 pre-dose to 24 hours post-dose (Day 2 in Part 1; Day 11 in Part 2)
  Mean absolute value
12-lead ECG parameters extracted from Holter (HR, PR, QRS, QTcF and QT) | From Day 1 pre-dose to 24 hours post-dose (Day 2 in Part 1; Day 11 in Part 2)
  Mean change from baseline
12-lead ECG parameters extracted from Holter (HR, PR, QRS, QTcF and QT) | From Day 1 pre-dose to 24 hours post-dose (Day 2 in Part 1; Day 11 in Part 2)
  Mean difference vs. placebo in change from baseline.
12-lead ECG parameters extracted from Holter (HR, PR, QRS, QTcF and QT) | From Day 1 pre-dose to 24 hours post-dose (Day 2 in Part 1; Day 11 in Part 2)
  The number and percentage of subjects with:
  * QTcF > 450 ms, > 480 ms and > 500 ms;
  * Change from baseline in QTcF > 30 ms and > 60 ms
12-lead Holter abnormal findings (total pauses > 2.5 seconds, atrial fibrillation and atrial flutter, ventricular runs, premature atrial contractions (PAC) burden, premature ventricular contractions (PVC) burden, other aberrant morphologies | From Day 1 pre-dose to 24 hours post-dose (Day 2 in Part 1; Day 11 in Part 2)
Mean 24-hour heart rate (HR0-24h, from 12-lead Holter recording) and mean hourly HR | From Day 1 pre-dose to 24 hours post-dose
Blood laboratory tests evaluation: chemistry, haematology | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Shift table will be presented by treatment at each post-dose time point
Blood laboratory tests evaluation: chemistry, haematology | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Mean absolute value will be presented by treatment
Blood laboratory tests evaluation: chemistry, haematology | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Mean change from baseline (Day -1) will be presented by treatment at each post-dose time point
Urine laboratory tests evaluation (urine strip): urinalysis | From Day 1 pre-dose to the first follow-up visit (15 ±3 days after Day 1 for Part 1; between 7 and 14 days after Day 10 for Part 2)
  Urinalysis values will be presented in the listings for each subject

SECONDARY OUTCOMES:
CHF6467 AUC0-24h | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Area under the concentration-time curve from time 0 to 24 h
CHF6467 AUC0-t | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Area Under the Curve from time 0 to time t
CHF6467 AUC0-∞ | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Area Under the Curve from time 0 Extrapolated to Infinity
CHF6467 Cmax | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Maximum Serum Concentration
CHF6467 tmax | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Time corresponding to maximum concentration
CHF6467 t½ | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Terminal half-life
CHF6467 CL/F | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Total body clearance
CHF6467 Vd/F | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
  Apparent volume of distribution
CHF6467 dose normalized AUC0-24h | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
CHF6467 dose normalized AUC0-t | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
CHF6467 dose normalized AUC0-∞ | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
CHF6467 dose normalized Cmax | From Day 1 pre-dose to the end of treatment (Day 1 in Part 1; Day 10 in Part 2)
CHF6467 concentration in Cerebrospinal fluid (CSF) | At either 1, 2, 4 or 6 hours post-dose on Day 1 (Part 1) or Day 10 (Part 2)
CHF6467 Antidrug Antibodies (ADA) detection in serum | From Day 1 pre-dose to last follow-up visit (29 ±3 days after Day 1 for Part 1; 85 ±3 days after Day 1 for Part 2)
CHF6467 Cmin | Post-dose on Day 9
  Minimum Serum Concentration
CHF6467 tmin | Post-dose on Day 9
  Time corresponding to minimum concentration
CHF6467 Cav | Post-dose on Day 9
  Average Serum Concentration
CHF6467 Rac Cmax | Comparison Day 9 vs Day 1
  Accumulation Ratio considering Cmax
CHF6467 Rac AUC0-24h | Comparison Day 9 vs Day 1
  Accumulation Ratio considering AUC0-24h

CONTACTS AND LOCATIONS:
Overall Officials: Maya Dabcheva, MD, Principal Investigator — MC Comac Medical Ltd.
Locations (1):
- Bulgaria MC Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No